CLINICAL TRIAL: NCT03536234
Title: A Prospective, Randomized, Open Study on the Efficacy and Safety of the GnRH Analogue Triptorelin for HIV-1 Reservoir Reduction in ART Treated HIV-1 Infected Patients
Brief Title: Efficacy and Safety of GnRH Analogue Triptorelin for HIV-1 Reservoir Reduction in ART Treated HIV-1 Infected Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immune System Regulation AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISR-003
Record Dates: First submitted 2018-04-20; First posted 2018-05-24 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triptorelin (GnRH analogue) (Experimental)
  Interventions: Drug: Triptorelin acetate depot
- Control group (No Intervention)

INTERVENTIONS:
Drug: Triptorelin acetate depot — 3.75 mg triptorelin depot (monthly injections). 3 doses in total
  Arms: Triptorelin (GnRH analogue)

SUMMARY:
An open, randomised, parallel arm phase IIa study. 52 HIV-1 infected patients will be randomised (in a 1:1 ratio) to either an active group or a control group. The active group will receive the GnRH analogue triptorelin depot monthly at baseline, week 4 and week 8. Patients in the active group and in the control group will continue their triple combination antiretroviral therapy (ART) during the study without changes; unless there is rationale for change on medical ground. In order to prevent the negative effects of a low testosterone level, patients in the active group will be offered to receive a single intramuscular depot injection of testosterone approximately 7 days after triptorelin treatment. This depot administration will keep the serum testosterone on a normal level until the next triptorelin dose. This will be repeated when triptorelin is administered at week 4 and week 8. Total study period is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male gender
2. 18 to 65 years of age, inclusive, at the time of informed consent
3. Ability and willingness to give a written or orally witnessed informed consent
4. HIV-1 infection as documented by HIV antibody test
5. CD4+ cell count >300 cells/μL at screening
6. Total HIV-1 DNA level between 100 to 5000 copies/million PBMC as measured by real-time PCR within 4 months prior to screening
7. Plasma HIV-1 RNA level <50 copies/mL for the last year (one blip allowed; blip defined as HIV RNA between 50-150 copies/mL) including a plasma HIV-1 RNA level <50 copies/mL at screening
8. On triple combination ART (two nucleoside reverse transcriptase inhibitors (NRTI) + one integrase inhibitor or protease inhibitor or one non-NRTI (NNRTI)) for minimum 36 months (assessed at screening)
9. Currently on continuous triple combination ART as specified above (i.e. no changes in medication) the past 4 months prior to screening

Exclusion Criteria:

1. Treatment failure while on triple ART
2. Nadir CD4+ count < 200 cells/μL
3. History of any immunodeficiency disease or condition other than HIV, chronic clinically significant illness or autoimmune disease
4. Known positive result of screening for hepatitis B (surface antigen positive or detectable HBV DNA levels in blood) or hepatitis C (HCV RNA positive). Patient treated for HCV and assessed as cured by treating physician is eligible for the study
5. Serious ongoing infection
6. Abnormal liver biochemical tests > 2 x upper limit of normal (ULN) of aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase (ALP)
7. Total testosterone, LH or FSH levels at screening assessed as clinically abnormal by the Investigator
8. Current treatment with testosterone
9. History of any clinically significant kidney disease as determined by the Investigator or eGFR < 60 mL/min/1.73 m2 at screening. (Patients on dolutegravir with an eGFR<60 may be verified for study inclusion by analysis of cystatin C that should then be assessed as normal by the Investigator in order for the patient to be eligible)
10. Diabetes mellitus or a fasting plasma blood glucose >7.0 mmol/L at screening
11. Intolerance or contraindication to injectable triptorelin
12. Vital signs, physical examination or lab results that exhibit evidence of acute illness
13. Known history of moderate or severe depression (see definitions in ICD-10) within the past 5 years
14. Any congenital or acquired prolongation of the QTc interval and use of any drugs that has been proven to prolong the QTc interval (Normal QTc interval defined as <450 msec)
15. Involvement in any other drug study within 30 days prior to this study entry
16. An increased PSA (Prostate Specific Antigen) value that is assessed as abnormal by the treating physician
17. Any medical condition that in the opinion of the Investigator would compromise the patient's ability to participate in the study
18. Investigator considers the patient unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline to week 12 in total HIV-1 DNA levels in CD4+ cells in the active group compared to the mean change in the control group. | Baseline to 12 weeks time point

SECONDARY OUTCOMES:
Mean change of the HLA class 1 expression from baseline to week 12 in the active group compared to the mean change in the control group | Baseline to 12 weeks time point
Mean change in the CD4+ T-cell counts from baseline to week 12 in the active group compared to the mean change in the control group. | Baseline to 12 weeks time point
Mean change in the CD8+ T-cell counts from baseline to week 12 in the active group compared to the mean change in the control group. | Baseline to 12 weeks time point
Number of adverse events in active group compared to control group | Baseline to 12 weeks time point
  Adverse events will be presented by Medical Dictionary for Regulatory Activities MedDRA) preferred term (PT) and system organ class (SOC).
Number and percentage of patients reporting any adverse events in active group compared to control group | Baseline to 12 weeks time point
  Number and percentage of patients reporting any adverse event will be be presented by MedDRA PT and SOC.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Winqvist, MD, PhD, Study Director — ISR AB
Locations (5):
- Germany (2):
  - Zentrum für Infektiologie Berlin Prenzlauer Berg, Berlin
  - MVZ Karlsplatz, Munich
- Sweden (3):
  - Östra sjukhuset, Gothenburg
  - Södersjukhuset, Stockholm
  - Karolinska University Hospital Huddinge, Stockholm